CLINICAL TRIAL: NCT04160689
Title: Influence of the Implant-Abutment Connection on the Ratio Between Height and Thickness of Tissues at the Buccal Implant Zenith: a Perspective Randomised 3d Comparative Analysis on 188 Implants
Brief Title: Influence of the Implant Connection on Facial Tissues Maturation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Marco Farronato, Principal Investigator, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Bone Loss; Periodontal Bone Loss; Implant Tissue Failure
MeSH Terms: conditions — Bone Diseases, Metabolic; Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Anyridge (Mega'Gen, Korea) 5° conical internal hexed connection
  Interventions: Biological: implantology
- Group 2 (Active Comparator): Core (Bioimplant, Italy) 35° conical internal hexed connection (screw-vent style)
  Interventions: Biological: implantology

INTERVENTIONS:
Biological: implantology — placing of implant

SUMMARY:
The substitution of a tooth with a fixture often induces undesired morphological changes, resulting in a deterioration of the aesthetic appearance. The purpose of this study is to compare the soft tissue behavior next to two different implant connections: 5° (group 1) and 35° hexed (group 2), conical, internal with switching platform design after 12 months of functional provisionalization

ELIGIBILITY:
Inclusion Criteria:

* Missing teeth
* good oral hygiene
* good systemic health

Exclusion Criteria:

* lactation
* pregnancy
* heavy smoking (more than 20 cigarettes/day)
* severe medical conditions that could affect periodontal health and peri-implant tissue response
* use of drugs correlated to periodontal hypertrophy
* bone volume that required bone augmentation procedures before implant placement as well as soft tissue graft or any kind of peri-implant tissue engineering

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
height of the peri-implant mucosa (MH) | after 12 months
  This measurement (MH) corresponds to the depth of the implant referred to the most coronal point of the buccal mucosa measured according to the main implant axis digitally calculated by 3D software Gom.
The width (MT) of the peri-implant mucosa | 12 months
  was calculated from the vestibular shoulder of the analogue to the external mucosa point perpendicular to the implant major axis digitally calculated by 3D software Gom.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farronato D, Pasini PM, Manfredini M, Scognamiglio C, Orsina AA, Farronato M. Influence of the implant-abutment connection on the ratio between height and thickness of tissues at the buccal zenith: a randomized controlled trial on 188 implants placed in 104 patients. BMC Oral Health. 2020 Feb 17;20(1):53. doi: 10.1186/s12903-020-1037-5. PMID 32066431